CLINICAL TRIAL: NCT02205073
Title: A RANDOMIZED, DOUBLE-BLIND, THREE PERIOD CROSS-OVER, PLACEBO CONTROLLED, PROOF OF MECHANISM STUDY TO INVESTIGATE THE EFFECT OF RG7314 ON VASOPRESSIN (AVP) PATHWAY ACTIVATION IN HEALTHY MALE SUBJECTS
Brief Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Crossover Study of RG7314 on the Potential Regulation of Higher Brain Functions in Healthy Male Participants: Proof of Mechanism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BP29412; 2014-000867-42 (EudraCT Number)
Record Dates: First submitted 2014-06-19; First posted 2014-07-31 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Dosing Period 1 (Placebo Comparator)
  Interventions: Drug: Placebo RD + Placebo SD
- Dosing Period 2 (Active Comparator)
  Interventions: Drug: Placebo RD + AVP SD
- Dosing Period 3 (Experimental)
  Interventions: Drug: RG7314 RD + AVP SD

INTERVENTIONS:
Drug: Placebo RD + AVP SD — Placebo (matching to study drug) repeat doses + intranasal AVP single dose
  Arms: Dosing Period 2
Drug: Placebo RD + Placebo SD — Placebo (matching to study drug) repeat doses + intranasal Placebo (matching to intranasal AVP) single dose
  Arms: Dosing Period 1
Drug: RG7314 RD + AVP SD — RG7314 repeat doses + intranasal AVP single dose
  Arms: Dosing Period 3

SUMMARY:
This is a single site, randomized, double-blind, three period cross-over, placebo-controlled, proof of mechanism study in healthy male subjects. The study will investigate whether the directionality of brain activity and connectivity in response to intranasal vasopressin treatment is similar to earlier studies and explores the effect of short-term treatment with RG7314 on functional MRI as a pharmacodynamic marker. While in the scanner, the participants will be asked to perform a face matching task and a Theory of Mind task, among other assessments. Participants' exposure to study drug will be assessed and all participants will receive follow-up examination 1 and 4 weeks after last dose.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed, healthy non-smoker male adults, 18 to 45 years of age
* A body mass index between 18 to 32 kg/m2 inclusive and total weight in the range of 50-100 kg
* Participants and their partners of childbearing potential must use 2 methods of contraception, one of which must be a barrier method for the duration of the study and for 90 days after the last dose
* In the investigator's opinion, the subject is deemed appropriate for participation in the study, capable of following the study schedule of assessments and complying with the study restrictions and discontinuation of prohibited medication will not pose undue risks to the participants

Exclusion Criteria:

* History of alcohol and/or substance abuse/dependence
* History of relapsing or current psychiatric or neurological disorders
* Participants who, in the Investigator's judgment, pose a suicidal risk, or any subject with a history of suicidal attempts or behavior
* Positive results for serology test for HIV, Hepatitis B, hepatitis C viruses
* Confirmed (e.g. 2 consecutive measurements) clinically significant abnormality on 12-lead electrocardiogram (ECG), including a QTcF of >/= 450 milliseconds
* Confirmed clinically significant abnormality in vital signs, clinical chemistry and/or urinalysis
* Active stomach ulcer disease or active gastrointestinal bleeding
* Personal or family history (first or second degree relatives) of cerebral aneurysm
* Personal history of stroke or traumatic head injury
* Confirmed clinically significant abnormality in parameters of hematology or coagulation
* History of coagulopathies, bleeding disorders or blood dyscrasias
* History of hematological malignancy or myelosuppression (including iatrogenic).
* Contraindications for MRI scans or any brain/head abnormalities restricting MRI eligibility
* Fulfillment of any of the MRI contraindications on the standard radiography screening questionnaire
* Use of prohibited medications within 2 weeks prior to randomization, or 5 half-lives (whichever is longer)
* Participation in an investigational drug study within 90 days prior to randomization
* Donation or loss of blood over 500 mL within three months prior to randomization
* Chronic rhinitis, allergic rhinitis, nasal polyps or any other nasal pathology that may affect the absorption of intranasal AVP according to investigator judgment
* Concomitant disease, condition or treatment which might interfere with the conduct of the study, or what would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Unwilling or unable to comply with the following lifestyle guidelines: (1) participants will abstain from alcohol for the entire study participation; (2) abstinence from any psychoactive agents or drugs of abuse for the duration of the study period; (3) participants should abstain from unusual strenuous exercise throughout the entire study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Replication of AVP-induced inhibition of anterior cingulate cortex (ACC) activity, as measured by BOLD fMRI during a face matching task, differences between treatments | After 6 days of dosing with RG7314/placebo and 40 - 130 minutes after application of intranasal vasopressin/placebo
Replication of AVP-induced inhibition of functional connectivity, as measured by BOLD fMRI during a face matching task, differences between treatments | After 6 days of dosing with RG7314/placebo and 40 - 130 minutes after application of intranasal vasopressin/placebo
Effect of RG7314 on the modulation of AVP pathway effects on ACC activity, as measured by BOLD fMRI during a face matching task, differences between treatments | After 6 days of dosing with RG7314/placebo and 40 - 130 minutes after application of intranasal vasopressin/placebo

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 12 weeks
Effect of RG7314 on brain activity modulated by AVP during an implicit and explicit emotional face processing task as evaluated by BOLD fMRI | After 6 days of dosing with RG7314/placebo and 40 - 130 minutes after application of intranasal vasopressin/placebo
Effect of RG7314 on brain activity modulated by AVP during a Theory of Mind task, as evaluated by BOLD fMRI | After 6 days of dosing with RG7314/placebo and 40 - 130 minutes after application of intranasal vasopressin/placebo
RG7314 plasma concentrations | 0h, 2:20h, 3h to 4:30h, 4:30h postdose on Days 6, 20, and 34

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Leiden, Netherlands